CLINICAL TRIAL: NCT03926286
Title: Fecal Microbial Transplant for Sjogrens Syndrome
Brief Title: Fecal Microbial Transplant (FMT) for Sjogrens Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Sjogrens Syndrome Foundation (Unknown); Microbiome Health Research Institute (Other)
Responsible Party: Principal Investigator, Anat Galor, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170733
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Sjogren's Syndrome
Keywords: Dry Eye; Auto-Immune Disorder
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMT for Sjogrens (Experimental): FMT- active ingredient coming from participant's screening stool
  Interventions: Drug: FMP-30

INTERVENTIONS:
Drug: FMP-30 — FMP-30 containing frozen human fecal microbiota administered as (3) units of FMP30 enema on Day 0 and Week1

SUMMARY:
This is an open label study to evaluate the effect of Fecal Microbiota Transplantation (FMT) on the gut microbiome and Systemic parameters.

ELIGIBILITY:
Inclusion criteria:

1. Positive diagnosis of Sjogrens syndrome, defined by meeting two or more of the following three criteria:

   * Positive serum anti-SS-A/Ro and/or anti-SS-B/La (or positive rheumatoid factor and ANA ≥ 1:320)
   * Labial salivary gland biopsy exhibiting focal lymphocytic sialadenitis with a focus score ≥ focus/4 mm2
   * Keratoconjunctivitis sicca with ocular staining score ≥ 3 (assuming that individual is not currently using daily eye drops for glaucoma, and has not had corneal surgery or cosmetic eyelid surgery in the last 5 years)

   Or by both of the following:

   Positive antibodies to one of the early markers of Sjogrens Syndrome:
   * Anti-salivary gland protein 1 (SP1)
   * Anti-carbonic anhydrase 6 (CA6)
   * Parotid secretory protein (PSP) Ocular staining score ≥ 3
2. Age ≥ 18 years at time of enrollment
3. Able to provide signed and dated informed consent
4. Women of child childbearing potential in sexual relationships with men must use an acceptable method of contraception§ from 30 days prior to enrollment until 4 weeks after completing study treatment.
5. Males must agree to avoid impregnation of women during and for four weeks after completing study treatment through use of an acceptable method of contraception*.

   * Includes, but is not limited to, barrier with additional spermicidal foam or jelly, intrauterine device, hormonal contraception (started at least 30 days prior to study enrollment), intercourse with men who underwent vasectomy.

     * Includes, but is not limited to, barrier with additional spermicidal foam or jelly and vasectomy.

Participant exclusion criteria

Exclusion Criteria:

1. Inability to provide informed consent and/or unable or unwilling to comply with protocol requirements.
2. Antibiotics for at least 2 weeks prior to FMT.
3. Active infection for >15 days: bacteremia, urinary tract infection, pneumonia or abdominal collection.
4. Known or suspected toxic megacolon and/or known small bowel ileus.
5. Previous FMT
6. Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy.
7. History of total colectomy or bariatric surgery.
8. Antibiotics for the treatment of an active infection or anticipated antibiotic use during trial duration.
9. Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy.
10. Expected life expectancy < 6 months
11. Patients with a history of severe anaphylactic or anaphylactoid food allergy.
12. Solid organ transplant patients ≤ 90 days post-transplant or on active treatment for rejection.
13. Neutropenia (<500 neutrophils/mL) or other severe immunosuppression. Patients on monoclonal antibodies to B and T cells, anti-tumor necrosis factor, glucocorticoids, antimetabolites, calcineurin inhibitors may be enrolled after consultation with their medical doctor.
14. Renal failure (GFR <30 or dialysis)
15. Human immunodeficiency virus+ controlled or not well controlled on antiretroviral therapy
16. Regular probiotic supplement use within prior 2 weeks to enrollment
17. Pregnancy or inability/unwillingness to use contraceptives.
18. A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study.
19. Exclusion on the discretion of the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with reported adverse events (AEs) and serious adverse events (SAEs) | 7 months
  As an evaluation of the safety of FMT, the number of participants with reported AEs and SAEs will be collected. All occurrences of AEs and SAEs, regardless of relatedness to FMT, will be reported and assessed by the clinician using the NIH CTCAE.
Number of participants with stable microbiome engraftment | month 3
  Engraftment will be analyzed via the Jensen-Shannon divergence (JSD). The engraftment scores will be the ratio between the donors and recipients at the bacterial genus level. Participants who successfully engraft will more closely resemble the donor microbial profile on JSD analysis.

SECONDARY OUTCOMES:
Change in dry eye symptoms | baseline, 1 week, 1 month, 3 months
  Dry eye symptoms will be measured by the Ocular Surface Disease Index (OSDI) Scale 0-100 Continuous with higher scores representing greater dry eye symptoms
Change in dry eye symptoms | baseline, 1 week, 1 month, 3 months
  Dry eye symptoms will be measured by the Dry Eye Questionnaire 5 (DEQ5) Scale Range 0-22 Continuous with a higher number representing greater symptomatology of dry eye
Change in diversity of bacterial communities | Pre FMT, 3 months post FMT
  This will be captured via high-throughput 16S gene sequencing using DNA extracted from stool specimens in study participants. The Shannon diversity index will be used as our primary measure of diversity.
Change in system immune profiles as measured by T cell populations | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  System immune profiles will be evaluated by completing a comprehensive immuno-phenotypic profile from blood samples evaluating T cell populations including Th1, Th17, and T regulatory cells.
Change in ocular and systemic symptoms as measured by the quality of life SF-12 Questionnaire | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  Ranges 0-100 with higher scores representing a better quality of life
Change in self-reported ocular pain as assessed by the Numerical Rating Scale(NRS) | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  NRS Scoring Ranges from 0-10 with 0=no pain sensation and 10=the most intense eye pain imaginable
Change in self-reported ocular pain as assessed by the Short-form McGill Pain Questionnaire(SFM-PQ) | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  SFM-PQ Scoring Ranges from 0-45 with zero to 45 with a higher score indicating more server eye pain
Change in self-reported ocular pain as assessed by the Neuropathic Pain Symptom Inventory (NPSI) | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  NPSI Scoring Ranges from 0-100 with the higher score indicating the worse pain imaginable.
Depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  PHQ-9 scoring Ranges from 0-27 with the higher score indicating a greater degree of depression
Depression as assessed by the Symptom Checklist 90 for Depression (SCL-90 Depression) | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  SCL-90 Depression scoring ranges from 0-4 with the higher score indicating a greater degree of depression.
Anxiety as assessed by the Symptom Checklist 90 for Anxiety (SCL-90 Anxiety) | Pre-FMT, 1 Week, 1 Month, 3 months post FMT
  SCL-90 Anxiety scoring ranges from 0-4 with the higher score indicating a greater degree of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Anat Galor, MD, MSPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaheer M, Wang C, Bian F, Yu Z, Hernandez H, de Souza RG, Simmons KT, Schady D, Swennes AG, Pflugfelder SC, Britton RA, de Paiva CS. Protective role of commensal bacteria in Sjogren Syndrome. J Autoimmun. 2018 Sep;93:45-56. doi: 10.1016/j.jaut.2018.06.004. Epub 2018 Jun 20. PMID 29934134
- [Background] De Luca F, Shoenfeld Y. The microbiome in autoimmune diseases. Clin Exp Immunol. 2019 Jan;195(1):74-85. doi: 10.1111/cei.13158. PMID 29920643
- [Background] Wang C, Zaheer M, Bian F, Quach D, Swennes AG, Britton RA, Pflugfelder SC, de Paiva CS. Sjogren-Like Lacrimal Keratoconjunctivitis in Germ-Free Mice. Int J Mol Sci. 2018 Feb 13;19(2):565. doi: 10.3390/ijms19020565. PMID 29438346
- [Background] de Paiva CS, Jones DB, Stern ME, Bian F, Moore QL, Corbiere S, Streckfus CF, Hutchinson DS, Ajami NJ, Petrosino JF, Pflugfelder SC. Altered Mucosal Microbiome Diversity and Disease Severity in Sjogren Syndrome. Sci Rep. 2016 Apr 18;6:23561. doi: 10.1038/srep23561. PMID 27087247